CLINICAL TRIAL: NCT02157649
Title: An Open-Label, Single-Dose, Crossover Comparative Bioavailability and Pharmacokinetic Study of Codeine Phosphate/Guaifenesin Extended-Release Tablet With Immediate-Release Tablet
Brief Title: Single Dose Trial of Extended Release Combination Tablet Codeine and Guaifenesin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nexgen Pharma, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: COGU506
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — Codeine; Guaifenesin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ER Tablet under Fasted Conditions (Experimental): Administration of a single dose of two ER Tablets, combination of Codeine/Guaifenesin 30gm/600mg, to subjects under fasted conditions.
  Interventions: Drug: ER Tablet under Fasted Conditions
- IR Tablet under Fasted conditions (Active Comparator): IR Tablet combination tablet of Codeine/Guaifenesin 20mg/400mg administered under fasted conditions as a single tablet every 4 hours during a 12 hour study [three doses]
  Interventions: Drug: IR Tablet under Fasted conditions
- ER Tablet under Fed Conditions (Experimental): Administration of a single dose of two ER Tablets, combination of Codeine/Guaifenesin 30gm/600mg, following a standard high-fat breakfast.
  Interventions: Drug: ER Tablet under Fed Conditions

INTERVENTIONS:
Drug: IR Tablet under Fasted conditions — Administration of IR Tablets combination of Codeine Phosphate/Guaifenesin 20mg/400mg every 4 hours for 12 hours total.
  Other Names: Codeine Phosphate/Guaifenesin 20mg/400mg
  Arms: IR Tablet under Fasted conditions
Drug: ER Tablet under Fed Conditions — Administration of two ER Tablet combination of Codeine Phosphate/Guaifenesin 30mg/600mg
  Other Names: Codeine Phosphate/Guaifenesin 30mg/600mg ER Tablet
  Arms: ER Tablet under Fed Conditions
Drug: ER Tablet under Fasted Conditions — Administration of two Codeine Phosphate/Guaifenesin 30mg/600mg ER Tablets under fasted conditions.
  Other Names: Codeine Phosphate/Guaifenesin 30mg/600mg ER Tablet
  Arms: ER Tablet under Fasted Conditions

SUMMARY:
The objectives of this study are (a) to determine if drug levels from a single dose of an extended-release Codeine/Guaifenesin tablet are similar to an immediate-release tablet given every four hours containing lower doses considered safe for over-the-counter use; (b) to evaluate if food affects the drug levels of this extended-release Codeine/Guaifenesin tablet after a single administration; and (c) to assess the safety and tolerability of the Codeine/Guaifenesin extended-release and immediate release tablet formulations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking volunteers (Female volunteers on a stable contraceptive medication regimen (> 3 months) may continue during the course of the study but its use must be documented), 18 to 45 years of age, inclusive; Ethnic Group: Arab & Mediterranean.
* Race: Mixed skin (white & black skin people).
* Body Mass Index (BMI) between 18 and 32 kg/m2, inclusive;
* willing and able to comply with the appropriate instructions necessary to complete the study, and;
* Fully informed of the risks of entering the study and willing to provide written informed consent.
* Subject is available for the whole study period and gave written informed consent
* If female, must be practicing abstinence or using a medically acceptable form of contraception (e.g., intrauterine device, hormonal birth control [continuously used for at least 3 months before first dose], or double barrier method). For the purpose of this study, all females are considered to be of childbearing potential unless they have been post - menopausal, biologically sterile, or surgically sterile (i.e., hysterectomy, bilateral oophorectomy, or tubal ligation) for more than one (1) yearNormal Physical examination.
* Vital signs within normal ranges.
* All laboratory screening results within the normal range, or being assessed as clinically Non-significant by the attending physician.
* Normal Kidney and Liver functions test.

Exclusion Criteria:

* Women of childbearing potential who don't use any contraceptive method, pregnant and/or lactating women.
* Ethnic Group (Non- Arab &/ or Non- Mediterranean)
* A significant abnormality in the pre-study physical examination that would place the volunteer at risk during participation in the trial;
* A clinical laboratory test value outside of the accepted reference range that is deemed by the Investigator to be clinically significant;
* Require prescription medication on a regular basis;
* A clinically significant illness during the 28 days prior to Period 1 dosing (as determined by the Investigator);
* History of serious illness that can impact fate of drugs
* History of gastrointestinal obstruction, constipation, inflammatory bowel disease, gallbladder disease, pancreas disorder over last 2 years, or recent (over last 3 years) gastrointestinal tract surgery, including gall bladder resection;
* Known history or presence of cardiac, pulmonary, endocrine, musculoskeletal, neurological, hematological or disease.
* Subjects with acute pulmonary insufficiency, respiratory depression, acute or chronic severe respiratory insufficiency or history of any of these
* History of head injury, seizures over last 4 years deemed by the Investigator to be clinically significant;
* Mental disease
* History of kidney disease or urination problem over last 2 years deemed by the Investigator to be clinically significant
* Subjects with renal and/or hepatic insufficiency should be excluded
* Presence of any significant physical or organ abnormality
* History of low blood pressure is deemed by the Investigator to be clinically significant;
* A positive Hepatitis B surface antigen, Hepatitis C antibody screen, or a reactive HIV antibody screen;
* Known or suspected hypersensitivities, allergies, or other contraindications to Codeine or a related opioid and/or Guaifenesin;
* History of severe allergy or allergic reactions to study drug or related drugs or heparin
* Known history or presence of food allergies, or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
* Known or suspected history of drug abuse within lifetime as judged by the Investigator;
* History of alcohol abuse or excessive intake of alcohol within last 5 years as judged by the Investigator;
* Positive screen for drugs of abuse, alcohol, or cotinine (nicotine) at screening or on admission to the unit prior to administration of investigational products;
* Use of drugs that induce or inhibit the hepatic metabolizing cytochrome P450 2D6 enzymes, within 30 days prior to administration of study formulations. Examples of inducers include: piperidins, carbamazepine, dexamethasone, rifampin. Examples of inhibitors include: cimetidine, diphenhydramine, fluvastatine, methadone, and ranitidine;
* Use of prescription medications within 21 days and OTC medications (including vitamins or herbal products) within 7 days (excluding flu vaccination) prior to the first administration of the study medication without Sponsor approval;
* Intake of Alcohol, caffeine, or xanthine beverages 16 hrs before each study drug administration.
* Use of any investigational drug within 30 days prior to first dosing;
* Use of any tobacco-containing product within 6 months of first dosing;
* Donated more than 400 mL of blood within 4 weeks before first dosing;
* Participation in another bioequivalence study and/or Clinical trials within 80 days prior to the start of this study Period I
* Exhausting physical exercise in the last 48 hours (e.g. weight lifting) or any recent significant change in dietary or exercise habits.
* Abnormal vital signs
* Abnormal Kidney and Liver functions test.
* In the opinion of the Investigator, unlikely or unable to successfully complete the study;
* Volunteer is vegetarian.
* Vomiting, Diarrhea on admission.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Serum Levels of Codeine and Guaifenesin | 20 samples over 24 hours
  Blood samples drawn prior to dosing with tablets, then at 19 additional time points over the next 24 hours.

SECONDARY OUTCOMES:
Safety and Tolerability | 24 hours
  Collect adverse event data during the dosing and sampling intervals

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaceutical Research Unit, Amman, Jordan